CLINICAL TRIAL: NCT00337675
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel-Group Study Evaluating the Effects of 2 Different Regimens of Montelukast (Daily Dosing and Intermittent, Episode-Driven Dosing) Compared With Placebo in the Treatment of Episodic Asthma in Children Aged 6 Months to 5 Years
Brief Title: Intermittent and Daily Dosing for Episodic (Periodic) Asthma (0476-302)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-302; MK0476-302; 2006_015
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm 1: drug + episodic supplemental placebo (Active Comparator): Montelukast once a day (qd) + episode driven supplemental placebo qd for 12 days for a 52-wk treatment period
  Interventions: Drug: montelukast sodium
- Arm 2: placebo comparator + episodic supplemental drug (Active Comparator): Placebo qd + episode driven supplemental Montelukast qd for 12 days for a 52-wk treatment period
  Interventions: Drug: montelukast sodium
- Arm 3: placebo comparator + episodic supplemental placebo (Placebo Comparator): Placebo qd + episode driven supplemental placebo qd for 12 days for a 52-wk treatment period
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 4 mg (or 5 mg, depending on age of patient) qd + episode driven supplemental Pbo qd for 12 days for a 52-wk treatment period.
  Other Names: MK0476; Singulair®
  Arms: Arm 1: drug + episodic supplemental placebo
Drug: Comparator: Placebo (unspecified) — Placebo (Pbo) qd + episode driven supplemental Pbo for 12 days for a 52-wk treatment period.
  Arms: Arm 3: placebo comparator + episodic supplemental placebo
Drug: montelukast sodium — Pbo qd + episode driven supplemental Montelukast 4 mg (or 5 mg, depending on age of patient) qd for 12 days for a 52-wk treatment period.
  Other Names: MK0476; Singulair®
  Arms: Arm 2: placebo comparator + episodic supplemental drug

SUMMARY:
This is a year-long study evaluating the efficacy of both daily and intermittent treatment of asthma in children who experience symptoms episodically (i.e., seasonally, usually in the context of upper respiratory tract infection).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 months to 5 years with episodic (periodic) asthma

Exclusion Criteria:

* Patients who are not in otherwise good health
* Patients who have persistent asthma (continual asthma symptoms)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1771 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valovirta E, Boza ML, Robertson CF, Verbruggen N, Smugar SS, Nelsen LM, Knorr BA, Reiss TF, Philip G, Gurner DM. Intermittent or daily montelukast versus placebo for episodic asthma in children. Ann Allergy Asthma Immunol. 2011 Jun;106(6):518-26. doi: 10.1016/j.anai.2011.01.017. Epub 2011 Mar 4. PMID 21624752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 111 centers worldwide.
  Patient screening began 16-Oct-2006 and the first patient was randomized on 3-Nov-2006.
  The last patient's last visit was completed on 12-Aug-2009.
Pre-assignment Details: 1979 screened; 208 excluded.
  Randomized patients met the following criteria: age 6-71 months, a history of episodic asthma symptoms that ranged between 2 and 6 episodes, depending on age, that were separated in time by periods without asthma symptoms. Patients had at least 1 corticosteroid treatment or were hospitalized for asthma at least 1 time.
Groups:
- Daily Montelukast: Patients were randomized to receive montelukast 4 mg (tablets or oral granules, depending on patient age) once daily at bedtime for 52 weeks plus intermittent 12-day courses of matching-image placebo (tablets or oral granules) once daily at bedtime (a course was initiated as needed for symptoms of imminent respiratory infection or episode of breathing problems) during the 52-week study period.
- Intermittent Montelukast: Patients were randomized to receive matching-image placebo to montelukast 4 mg (tablets or oral granules, depending on age) once daily at bedtime for 52 weeks plus intermittent 12-day courses of montelukast 4 mg (tablets or oral granules) once daily at bedtime (a course was initiated as needed for symptoms of imminent respiratory infection or episode of breathing problems) during the 52-week study period.
- Placebo: Patients were randomized to receive matching-image placebo to montelukast 4 mg (tablets or oral granules, depending on age) once daily at bedtime for 52 weeks plus intermittent 12-day courses of matching-image placebo (tablets or oral granules) once daily at bedtime (a course was initiated as needed for symptoms of imminent respiratory infection or episode of breathing problems) during the 52-week study period.
Period: Overall Study
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo
Started | 589 | 591 | 591
Completed | 492 | 488 | 492
Not Completed | 97 | 103 | 99
Not completed — Adverse Event | 10 | 9 | 19
Not completed — Lack of Efficacy | 10 | 7 | 9
Not completed — Lost to Follow-up | 22 | 19 | 17
Not completed — Physician Decision | 9 | 17 | 14
Not completed — Protocol Violation | 21 | 24 | 19
Not completed — Withdrawal by Subject | 25 | 25 | 19
Not completed — Progressive Disease | 0 | 2 | 0
Not completed — Trial Terminated | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo | Total
Number analyzed (Participants) | 589 | 591 | 591 | 1771
Age, Continuous [Mean (Full Range); unit: Months] | 39.0 [6.0 to 71.0] | 39.5 [6.0 to 71.0] | 39.3 [7.0 to 71.0] | 39.2 [6.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 226 | 238 | 703
  Male | 350 | 365 | 353 | 1068

OUTCOME MEASURES:

1. Primary Outcome: Number of Asthma Episodes Culminating in Asthma Attack Over the 1-year Treatment Period
Description: The rate per year of asthma episodes culminating in an asthma attack for each of the 3 treatment groups. Asthma attacks were defined as respiratory symptoms requiring healthcare resource utilization (HRU), which comprised unscheduled visits to a physician or emergency department, treatment with corticosteroids (oral, rectal, or inhaled), or hospitalization. Each day during an episode, the patient's legal guardian recorded all the HRU that was required specifically for breathing problems.
Time Frame: 1-year treatment period
Population: Full Analysis Set (FAS): all randomized patients who took at least one dose of blinded study drug. Of 1771 patients randomized, 5 never took study drug and 9 were not included due to Good Clinical Practice compliance concerns. Therefore, 1757 patients were included in the FAS population.
Measure: Mean (95% Confidence Interval); unit: Asthma attacks within episodes per year
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo
Number analyzed (Participants) | 584 | 588 | 585
Asthma attacks within episodes per year | 0.99 [0.86 to 1.14] | 1.06 [0.92 to 1.22] | 1.05 [0.92 to 1.20]
Statistical Analysis 1: Comparison: Daily Montelukast vs Placebo; The primary hypothesis stated that montelukast (daily regimen, or [intermittent and daily regimens]), compared with placebo, results in a decrease in the number of asthma episodes culminating in asthma attack in pediatric patients aged 6 months to 5 years with episodic asthma and treated over 1 year. A sample size of 450 evaluable patients per arm allowed the detection of a difference in rate of 23% with 90% power; Test type: Superiority or Other; p = 0.510, Regression, Poisson — Multiplicity adjustment across regimens was addressed through step-down testing. Daily montelukast versus placebo was tested first; if this comparison was significant, intermittent montelukast versus placebo was tested. The significance level was 5%; A Poisson regression model containing factors for treatment, age group, and geographic region, and an offset for number of days in study was used; Rate reduction = 5.3, 95% CI [-11.4 to 19.6], Standard Error of Mean 7.3 — Rate reduction = (1 - montelukast-adjusted annual rate/placebo-adjusted annual rate) x 100%
Statistical Analysis 2: Comparison: Intermittent Montelukast vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.884, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Rate reduction = -1.2, 95% CI [-19.2 to 14.0], Standard Error of Mean 7.8 — Rate reduction = (1 - montelukast-adjusted annual rate/placebo-adjusted annual rate) x 100%

2. Secondary Outcome: Daily Average of Wheeze and Difficulty Breathing in the 3 Days Prior to Start of an Asthma Attack Within an Asthma Episode
Description: Each day during an asthma episode, the patient's legal guardian was asked to rate each of the symptoms of wheeze and difficulty breathing on a 6-point scale (Scale 0 (best) to 5 (worst)). The average of the individual symptom scores on each of the 3 days prior to an asthma attack was reported. If a patient had multiple episodes during 1 year, the symptom scores were averaged across all the episodes.
Time Frame: 1 Year
Population: Only patients who experienced an asthma attack within an episode and did not start their intermittent study medication on the day of the attack could be included. Therefore, a total of 452 patients were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo
Number analyzed (Participants) | 138 | 162 | 152
Units on a Scale | 1.69 [1.49 to 1.88] | 1.70 [1.52 to 1.89] | 1.88 [1.69 to 2.07]
Statistical Analysis 1: Comparison: Daily Montelukast vs Placebo; The secondary hypothesis stated that montelukast (daily regimen, or [intermittent and daily regimens]), compared with placebo, results in improvement of respiratory symptoms assessed over 3 days prior to asthma attacks, or assessed over the 12-day treatment period of asthma episodes in pediatric patients aged 6 months to 5 years with episodic asthma and treated over 1 year; Test type: Superiority or Other; p = 0.176, ANOVA — Multiplicity adjustment across regimens and across primary and secondary endpoints was addressed through step-down testing. Within the 2 endpoints assessing severity, adjustment for multiplicity was performed using Hochberg's method; An ANOVA model containing factors for treatment, age group, and geographical region was used; Least-Squares Mean Difference = -0.19, 95% CI [-0.46 to 0.09], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Intermittent Montelukast vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.202, ANOVA — [p-value comment as in outcome 2, analysis 1]; An ANOVA model containing factors for treatment, age group, and geographical region was used; Least-Squares Mean Difference = -0.17, 95% CI [-0.44 to 0.09], Standard Error of Mean 0.14

3. Secondary Outcome: Daily Average of the Mean Symptom Scores (Wheeze, Difficulty Breathing, Interference With Activity, and Daytime Cough) Assessed Over the 12-day Treatment Period of Asthma Episodes
Description: Each day during an asthma episode, the patient's legal guardian was asked to rate each of the symptoms of Wheeze, Difficulty Breathing, Interference with Activity, and Daytime Cough on a 6-point scale (Scale 0 (best) to 5 (worst)). The average of the individual symptom scores on each of the 12 days of intermittent treatment for an episode (before the first attack) was reported. If a patient had multiple episodes over 1 year, the symptom scores were averaged across all the episodes.
Time Frame: 1 Year
Population: Patients with at least one episode culminating in an attack were included; therefore, 1120 patients were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo
Number analyzed (Participants) | 365 | 387 | 368
Units on a Scale | 1.08 [1.00 to 1.16] | 1.09 [1.01 to 1.17] | 1.20 [1.12 to 1.28]
Statistical Analysis 1: Comparison: Daily Montelukast vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.045, ANOVA — Multiplicity adjustment across regimens and across primary and secondary endpoints was addressed through step-down testing. Within the family of secondary endpoints, adjustment for multiplicity was performed using Hochberg's method; An ANOVA model containing factors for treatment, age group, and geographical region was used; Least-Squares Mean Difference = -0.12, 95% CI [-0.24 to 0.00], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intermittent Montelukast vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.061, ANOVA — [p-value comment as in outcome 3, analysis 1]; An ANOVA model containing factors for treatment, age group, and geographical region was used; Least-Squares Mean Difference = -0.11, 95% CI [-0.23 to 0.00], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: October 2006 through August 2009
Arm/Group | Daily Montelukast | Intermittent Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 28/584 | 41/588 | 33/585
Other Adverse Events (participants affected / at risk) | 481/584 | 506/588 | 486/585
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Montelukast (N=584) | Intermittent Montelukast (N=588) | Placebo (N=585)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Adenoiditis (Infections and infestations) | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Kawasaki's disease (Infections and infestations) | 1 | 0 | 0
Laryngotracheitis obstructive (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Parotid abscess (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4 | 4
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Immune system disorders) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Varicella (Infections and infestations) | 0 | 1 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1
Viral rash (Infections and infestations) | 1 | 0 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 17 | 14
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Montelukast (N=584) | Intermittent Montelukast (N=588) | Placebo (N=585)
Diarrhoea (Gastrointestinal disorders) | 35 | 49 | 43
Vomiting (Gastrointestinal disorders) | 22 | 31 | 30
Pyrexia (General disorders) | 94 | 87 | 80
Bronchitis (Infections and infestations) | 33 | 40 | 32
Influenza (Infections and infestations) | 30 | 31 | 27
Nasopharyngitis (Infections and infestations) | 110 | 110 | 81
Otitis media (Infections and infestations) | 44 | 55 | 45
Pharyngitis (Infections and infestations) | 59 | 64 | 67
Rhinitis (Infections and infestations) | 36 | 33 | 30
Sinusitis (Infections and infestations) | 39 | 49 | 27
Tonsillitis (Infections and infestations) | 38 | 42 | 37
Upper respiratory tract infection (Infections and infestations) | 81 | 76 | 82
Varicella (Infections and infestations) | 36 | 15 | 28
Asthma (Respiratory, thoracic and mediastinal disorders) | 332 | 338 | 319
Cough (Respiratory, thoracic and mediastinal disorders) | 91 | 101 | 93
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 46 | 44 | 31
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 29 | 29
Wheezing (Respiratory, thoracic and mediastinal disorders) | 33 | 31 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.